CLINICAL TRIAL: NCT01193036
Title: Symptom Burden in Patients With Cancer- and Treatment-Related Skin Problems
Status: Terminated | Type: Observational
Why Stopped: Low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-0551
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Skin Cancer
Keywords: Psychosocial; Skin Problems; Supportive Care; Melanoma; Questionnaire
MeSH Terms: conditions — Skin Neoplasms; Melanoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Interview
  Interventions: Behavioral: Part 1: Interview + Questionnaires
- Symptom Inventory Assessment
  Interventions: Behavioral: Part 2: Multiple Questionnaires

INTERVENTIONS:
Behavioral: Part 1: Interview + Questionnaires — Questionnaires to be completed immediately after interview, which will take approximately 15 minutes.
  Groups: Interview
Behavioral: Part 2: Multiple Questionnaires — Questionnaires to be repeated about every 2 weeks for 1 year.
  Groups: Symptom Inventory Assessment

SUMMARY:
Objectives:

The objective of this study is to develop a valid and reliable measure of the symptom burden experienced by patients with cancer experiencing disease-related skin problems and to delineate this burden over time.

The Primary Aim is to develop and validate an M.D. Anderson Symptom Inventory (MDASI) module (the MDASI-Derm), compliant with FDA standards for patient-reported outcomes (PROs), to measure the severity of multiple symptoms and the impact of these symptoms on daily functioning in patients with cancer-related skin problems. We hypothesize that the MDASI-Derm will be valid and reliable for measuring the severity of multiple symptoms and the impact of these symptoms on daily functioning in patients with cancer-related skin problems.

The Secondary Aims are:

1. to develop a detailed description of the severity and interference with daily activities of symptoms experienced by patients with cancer-related skin problems;
2. to assess the impact of symptom severity on standard function and quality of life (QOL) measures including both quantitative (Eastern Cooperative Oncology Group [ECOG] Performance Status, single-item QOL, and Skindex-16 scales) and qualitative measures (patient interviews);
3. to evaluate the MDASI-Derm as an estimate of functional status and QOL in patients with cancer-related skin problems;
4. to identify common clusters of symptoms and symptom patterns occurring over multiple measurement time points in patients with cancer-related skin problems;
5. to define the qualitative symptom experience of patients with cancer-related skin problems;
6. to explore the feasibility of the Interactive Voice Response (IVR) system in measuring symptom severity and interference with daily activities over time in patients with cancer-related skin problems.

DETAILED DESCRIPTION:
Part I:

Interview:

If you agree to take part in this study, while you are at the clinic for a visit, you will be interviewed about skin problems and other symptoms that you have had since you began experiencing skin problems. The interview should take about 30 minutes to complete.

Part I:

Questionnaires:

After the interview, you will be asked to answer a general symptom questionnaire, a quality-of-life questionnaire, a skin-specific questionnaire, and some demographic questions (such as your age and marital status). It should take about 15 minutes to complete all 4 questionnaires.

Part II:

Symptom Questionnaires:

If you agree to take part in this study, you will complete a questionnaire about skin problems and other symptoms you are having. This symptom questionnaire will ask you to rate how severe your skin problems and other symptoms are and how the skin problems and other symptoms affect the activities of your daily life. It should take about 5 minutes to complete. You will complete the questionnaire at a routine clinic visit every 2 weeks for 1 year. If you do not have a clinic visit every 2 weeks, you will be called by an automated phone system so you may complete the questionnaire at least 1 time every 2 weeks.

You can decide what time is most convenient for the automated phone system to call you. If you are not available when the automated system calls, it will call you again at a later time. You will be given a secure user name and identification number to use with the automated phone system. The study staff will teach you how to use the automated phone system.

Two (2) days after you begin the study, you will fill out the symptom questionnaire again. You will take home a paper copy of the questionnaire with you from the clinic with a pre-addressed, stamped envelope given to you by the research staff so you can return it. The research staff will also ask for your telephone number so that they may contact you and remind you to complete the questionnaire.

Quality-of-Life/Demographic Questionnaires:

At the first visit, you will also be asked some demographic questions (such as your age and employment status). Answering these questions should take about 1 minute. Some of these questions (such as employment status) will be repeated at regular clinic visits. You will not be asked to do this more often than every 3-5 weeks.

At the first visit and at regular clinic visits, you will also rate your overall quality-of-life. This should take about 1 minute to complete. You will not be asked to do this more often than every 3-5 weeks.

At the first visit and at regular clinic visits, you will be asked to complete a second questionnaire that asks specific questions about how problems with your skin affect the quality of your life. This should take about 5 minutes to complete. You will not be asked to do this more often than every 3-5 weeks.

Opinion Questionnaire:

If you are 1 of the first 20 participants enrolled in Part 2 of this study, you will be asked questions about your opinion of the symptom questionnaire after you have completed it for the first time. For example, you will be asked if the symptom questionnaire was easy to understand and complete, and if there were any other questions that should be included. The study staff will use your opinion to decide if changes should be made to the questionnaire or if important symptom questions are missing from the questionnaire. This questionnaire should take about 5 minutes to complete.

Part I:

Length of Study:

After you have completed the interview and questionnaires, your participation on this study will be over.

Part II:

Length of Study You will be on study for 1 year. You will be off study after you complete the last symptom questionnaire.

This is an investigational study. Up to 60 participants will take part in this study. Up to 20 will be enrolled in Part 1 of this study. Up to 40 participants will be enrolled in Part 2 of this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Ability to read and speak English
3. Receiving treatment and/or follow up at M. D. Anderson Cancer Center
4. Residing where IVR service is available (Validation part of study only)
5. Rating of skin problem at its worse in the last 24-hours of at least 1 on a 0 to 10 scale where 0 is no skin problem and 10 is the skin problem as bad as can be imagined
6. Written consent to participate

Exclusion Criteria:

1. Medical condition (impaired speech that would preclude taking part in a 30 minute interview, deafness that would impair the ability to use the IVR system) or impaired performance status that would preclude participation in the study
2. Diagnosis of active psychosis or severe cognitive impairment as determined by physician
3. Active treatment (systemic drug therapy or radiation therapy) for a second malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Hospital and the Melanoma and Skin Center
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Severity of Multiple Symptoms/Impact of Symptoms on Daily Functioning | 1 year
  MDASI-Derm measure of severity + impact of 13 cancer-related core symptoms that cause most interference with daily activities; Severity of symptoms rated (with amount of interference with daily living) on scales from 0 to 10, with 0 meaning no symptom or interference and 10 meaning as severe or complete interference.

CONTACTS AND LOCATIONS:
Overall Officials: Loretta A. Williams, PhD, MSN, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org